CLINICAL TRIAL: NCT06733766
Title: Ultrasound-guided Thermal Ablation for Recurrent Thyroid Cancer: A Multicenter Study
Brief Title: Ultrasound-guided Thermal Ablation for Recurrent Thyroid Cancer
Status: Recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yu-kun Luo, Clinical Professor, Chinese PLA General Hospital
Other Study IDs: 2024-657
Record Dates: First submitted 2024-12-07; First posted 2024-12-13 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Recurrent Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ultrasound-guided thermal ablation: ultrasound-guided thermal ablation
  Interventions: Procedure: ultrasound-guided thermal ablation

INTERVENTIONS:
Procedure: ultrasound-guided thermal ablation — microwave ablation, radiofrequency ablation, laser ablation

SUMMARY:
To evaluate the long-term outcomes of ultrasound-guided thermal ablation for recurrent thyroid cancer

DETAILED DESCRIPTION:
To evaluate and predict the long-term outcomes of ultrasound-guided thermal ablation for recurrent thyroid cancer by a multicenter study

ELIGIBILITY:
Inclusion Criteria:

1. patient received thyroidectomy for thyroid cancer
2. recurrent lesions were pathologically proven to be malignant by core-needle biopsy or fine needle aspiration
3. no evidence of distant metastases.
4. follow-up period ≥12 months

Exclusion Criteria:

1. coagulation disorder, serious heart, respiratory, liver, or renal failure
2. dysfunction of the vocal cord on the opposite side

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with recurrent thyroid cancer
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
rate of disease progression | through study completion, an average of 6 months
  cervical lymph node metastases and persistent tumors confirmed by pathology, Distant metastasis detected by CT, positron emission tomography, or bone scan if there were suspicious symptoms.

SECONDARY OUTCOMES:
rate of complications | 1 week
  complication of ablation
rate of volume reduction | through study completion, an average of 6 months
  volume reduction of tumor after ablation on ultrasound and contrast-enhanced ultrasound
rate of tumor disappearance | through study completion, an average of 6 months
  complete disappearance of ablated tumor on ultrasound and contrast-enhanced ultrasound
Tg level | through study completion, an average of 6 months
  serum thyroglobulin level
rate of delayed surgery | through study completion, an average of 1 year
  patients underwent surgery after ablation because of anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Yukun Luo, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No